CLINICAL TRIAL: NCT04687800
Title: A Randomized, Clinical Investigation of the Dextenza 0.4mg Intracanalicular Insert Delivery System Used in Conjunction With Cataract Surgery Performed in Combination With Minimally Invasive Glaucoma Surgery
Brief Title: Clinical Investigation of the Dextenza 0.4mg Intracanalicular Insert Delivery System Used in Cataract Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to enroll due to lack of access to the Ambulatory Surgery Center.
Sponsor: Cathleen McCabe MD (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Cathleen McCabe MD, Principal Investigator, The Eye Associates
Organization: The Eye Associates (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The McTENZA Study
Record Dates: First submitted 2020-12-08; First posted 2020-12-29 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate; difluprednate

STUDY DESIGN:
Intervention Model Description: Open label prospective randomized comparative investigator -initiated study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza 0.4mg (Experimental): Intracanalicular insert
  Interventions: Drug: Dextenza 0.4mg intracanalicular Insert
- Durezol 0.05% (Active Comparator): difluprednate ophthalmic emulsion
  Interventions: Drug: Durezol 0.05% Ophthalmic Emulsion

INTERVENTIONS:
Drug: Dextenza 0.4mg intracanalicular Insert — intracanalicular insert delivery system
  Other Names: dexamethasone ophthalmic insert
  Arms: Dextenza 0.4mg
Drug: Durezol 0.05% Ophthalmic Emulsion — Standard therapy, topical steroid drop
  Other Names: difluprednate ophthalmic
  Arms: Durezol 0.05%

SUMMARY:
To monitor intraocular pressure in glaucoma patients after cataract surgery preformed in conjunction with minimally invasive glaucoma surgery (MIGS)

DETAILED DESCRIPTION:
The purpose of this study is to monitor glaucoma patients intraocular pressure (IOP) after cataract surgery performed in conjunction with minimally invasive glaucoma surgery. After qualifying for this study, subjects will be randomized in a 1:1 allocation of one of two arms. The purpose of this study is to determine if Dextenza (dexamethasone) 0.4mg intracanalicular insert delivery system, provides a decreased risk of elevated post-operative IOP vs. standard therapy controlled topical steroid Durezol (Difluprednate ophthalmic emulsion) 0.05%

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or Older
* Mild-to-moderate primary open angle glaucoma and visually significant cataract with plans to undergo clear cornea cataract surgery with Phacoemulsification and implantation of posterior chamber IOL combined with minimally invasive glaucoma surgery ( MIGS) procedure in both eyes.

Exclusion Criteria:

* Use of Topical steroid, systemic steroid or intravitreal steroid implants within last 3 months
* Previous Corneal surgery or pathology
* Active or history of chronic or recurrent inflammatory eye disease in either eye
* Ocular Pain in either eye
* Proliferative diabetic retinopathy in either eye
* Significant macular pathology detected on macular optical coherence tomography evaluation at the screening visit in either eye.
* Laser or incisional ocular surgery during the study period and 6 months prior in either eye
* Systemic concomitant pain medication management with the pharmacology class of Oxycodone
* Systemic NSAIDS use >/=750 mg daily
* Clinically significant macular edema
* History of cystoid macular edema in either eye

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure from Baseline | 30 days - IOP measured at day 1, day 14 and day 30
  Sustained tapered release of Dextenza compared to Durezol 4 week taper as measured by mean IOP from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen M McCabe, MD, Principal Investigator — The Eye Associates of Manatee
Locations (1):
- The Eye Associates of Manatee, Bradenton, Florida, United States

REFERENCES:
- See also: Sponsor/ site website — https://www.theeyeassociates.com/